CLINICAL TRIAL: NCT04508192
Title: Strength Effects of the Copenhagen Adduction Exercise Vs an Adductor Squeeze Exercise in Male Soccer Players
Brief Title: Copenhagen Adduction Exercise Vs an Adductor Squeeze Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Principal Investigator, Andreas Serner, Clinical Research Scientist, Aspetar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CAvsSQ
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Groin Injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomisation will be performed after baseline strength testing. Participants will be individually randomized to perform either the CA or the SQ exercise protocol. The randomisation sequence will be obtained using an online software (e.g. randomizer.org), and sealed, opaque envelopes containing group allocation will be prepared by an independent person not otherwise involved in the study, and who will be unaware of the baseline strength test results. All participants will be instructed not to perform any additional adductor exercise other than their allocated exercise and to keep their regular training as usual.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person performing the strength tests will be blinded to group allocation, and participants will be instructed not to reveal any information about their group allocation. In addition, the physiotherapist supervising the intervention procedures will not be allowed to know the results of the strength measurements of each player.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Copenhagen Adduction (Experimental): The CA is a high-intensity partner exercise where the player is lying on their side using the elbow of the lower forearm to support their body and the other arm placed along their body. The upper arm is supported by the partner who places their one hand under the knee and the other under the ankle, holding the leg approximately in the height of their hip. The player performs a 3-second concentric movement lifting their body until it reaches a straight line. At the same time, the other leg is adducted so that it touches the other leg. A 3-second eccentric adduction then follows with the body lowered halfway to the ground and the foot of the lower leg touching the ground without supporting the body.
  Interventions: Other: Exercise
- Adductor Squeeze (Active Comparator): The SQ exercise is an isometric hip adduction exercise with the player holding a ball between their knees. The player lies supine with the ball placed between the knees with the knees and hips flexed and the feet flat on the surface with the first toe is pointed straight forward.the player is asked to press against the ball as hard as they can The contraction is held for 10 seconds
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both interventions are simple strength exercises without technical equipment

SUMMARY:
The study aims to compare the effects of two different adduction exercises on adduction strength. Young male football players will be individually randomized to perform one of these exercises in addition to their normal training. The two exercise protocols are of 8 weeks duration and are matched in terms of total load.

DETAILED DESCRIPTION:
Methods Participants Male football players 16 years or older, who are participating in full team training in Greece, will be included in the study. The study will be conducted pre-season. During that time each player will have at least 4 training sessions and 1 match per week.

Exclusion criteria were

* any systematic resistance training of the hip adductors (> 1/week) in the preceding 1 month before study initiation.
* groin pain resulting in loss of one or more football matches/training sessions in the preceding 1 month prior to study initiation.
* any longstanding injury (≥ 6 weeks) in the lower extremities or in the hip/groin in the preceding 6 months prior to study initiation.
* pain of more than 2/10 on a numeric rating scale (NRS) when performing the adduction strength tests or exercises were also excluded.
* For analysis, players will be excluded if there was an adherence of less than 75% of the exercise sessions.

Ethics Ethical approval was obtained from University of West Attica ethics committee and all players will give their informed consent prior to inclusion in accordance with the Declaration of Helsinki.

Randomisation Randomisation will be performed after baseline strength testing. Participants will be individually randomized to perform either the CA or the SQ exercise protocol. The randomisation sequence will be obtained using an online software (e.g. randomizer.org), and sealed, opaque envelopes containing group allocation will be prepared by an independent person not otherwise involved in the study, and who will be unaware of the baseline strength test results. All participants will be instructed not to perform any additional adductor exercise other than their allocated exercise and to keep their regular training as usual.

Blinding The person performing the strength tests will be blinded to group allocation, and participants will be instructed not to reveal any information about their group allocation. In addition, the physiotherapist supervising the intervention procedures will not be allowed to know the results of the strength measurements of each player.

Training intervention Both groups will perform an 8-week training protocol with either the CA or the SQ exercise performed before or after the normal football training sessions.

Copenhagen Adduction exercise The CA is a high-intensity partner exercise where the player is lying on their side using the elbow of the lower forearm to support their body and the other arm placed along their body. The upper arm is supported by the partner who places their one hand under the knee and the other under the ankle, holding the leg approximately in the height of their hip. The player performs a 3-second concentric movement lifting their body until it reaches a straight line. At the same time, the other leg is adducted so that it touches the other leg. A 3-second eccentric adduction then follows with the body lowered halfway to the ground and the foot of the lower leg touching the ground without supporting the body. To ensure a correct performance the therapist instructs the players that there should not be any side flexion of the trunk or hip during the exercise. Each player performs one set on each side and then the players change roles. Each couple will be comprised of players of similar height and weight to ensure optimal conditions.

Adductor Squeeze exercise The SQ exercise is an isometric hip adduction exercise with the player holding a ball between their knees. The player lies supine with the ball placed between the knees with the knees and hips flexed and the feet flat on the surface with the first toe is pointed straight forward. Then the player is asked to press against the ball as hard as they can. The contraction is held for 10 seconds.

Load progression The CA will be performed with increasing number of repetitions during the intervention period as the only load progression variable. The number of sets will be kept at 2 sets per side throughout the study. Additionally, the total time under tension (TUT) of the CA protocol is adjusted to that of the SQ exercise. The SQ exercise has previously been suggested to be performed in two positions with 5 repetitions of 10 seconds each. This study will use only one exercise position for comparison, the SQ exercise will be performed for 10 repetitions.

Outcome measures The primary outcome measure of the study will be maximal eccentric adduction strength (EHAD). Secondary outcome measures will be maximal unilateral isometric adduction strength (IHAD), and DOMS. The distance between anterior superior iliac spine (ASIS) and the point of the handheld dynamometer placement will be measured to calculate torque (Nm/kg). Both the side-lying eccentric adduction and unilateral supine isometric strength measurements will be conducted on the dominant as well as non-dominant limb. Testing will be conducted in the club's training facility. The tester will use a handheld dynamometer following standardized procedures which have been shown to have a good intra-tester reliability: eccentric adduction strength ICC 0.91 (0.70-0.98), SEM: 6.3% and isometric adduction strength ICC 0.78 (0.30-0.95), SEM: 7.3%

Compliance Compliance and perceived loading will be recorded after every training session with the respective intervention exercise, while hip adductor DOMS will be recorded in respect of the previous training session. Perceived loading will be defined via the Borg CR10 scale and DOMS via a numerical ranking scale (NRS 0-10). All players will be instructed to avoid any type of training 24h before baseline and follow-up testing. Moreover, the follow-up testing will be conducted 3 days after the intervention to avoid DOMS potentially influencing the measures.

Statistical analyses Baseline and follow-up values as well as anthropometric data will be presented as mean SD, unless otherwise stated. A mixed analysis of variance (ANOVA) will be used to assess the interactions between groups (CA vs SQ) and time (baseline vs follow-up) on the dependent variables (EHAD, IHAD and DOMS). Additionally, the simple main effect of time will be analyzed using a dependent t-test. Cohen's d will be used for effect size (ES) calculation and will be set as small (0.2), moderate (0.5) and large (0.8) . Statistical significance level will be set at p 0.05. The data analysis will be performed using SPSS Statistics (v 26, IBM Corporation).

Sample size A sample size calculation was performed prior to study initiation using G*power software (v. 3.1, Heinrich-Heine-Universität, Düsseldorf, Germany). Based on previous studies the expected mean normalized eccentric adduction strength was set at 3.0 Nm/kg with a standard deviation (SD) of 0.6 Nm/kg. The minimal relevant difference in EHAD strength between groups was chosen to be 20%, and correlation was arbitrarily set at 0.5. With 80% power and a type-1 error risk of 5%, and a correlation a total sample size of 42 participants was adequate to detect a large moderate effect size. To account for dropouts during the intervention a minimum of 60 participants are included.

ELIGIBILITY:
Inclusion Criteria:

* Male football players 16 years or older, who were participating in full team training in Greece.

Exclusion Criteria:

* any systematic resistance training of the hip adductors (> 1/week) in the preceding 1 month before study initiation.
* groin pain resulting in loss of one or more football matches/training sessions in the preceding 1 month prior to study initiation.
* any longstanding injury (≥ 6 weeks) in the lower extremities or in the hip/groin in the preceding 6 months prior to study initiation.
* pain of more than 2/10 on a numeric rating scale (NRS) when performing the adduction strength tests or exercises were also excluded.
* For analysis, players will be excluded if there was an adherence of less than 75% of the exercise sessions.

Ages: 16 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Eccentric hip adductor strength | Change from baseline eccentric adductor strength at 8 weeks
  The athlete lies on the side of the tested leg with their hip and knee in a straight position. The hip and knee of the other leg are placed in 90deg of flexion with the knee placed on a box to maintain position of the pelvis. The athlete holds on to the side of the bed with one hand for stabilization. The examiner lifts the tested leg off the bed into full adduction and applies a downward force to the limb holding the HHD 5cm above the medial, while the athlete is asked to resist that force performing hip adduction "as hard as possible" Then the tester breaks the athlete's resistance applying a downward force. The procedure is performed three times with a 30-second rest between each of them and the highest value is recorded.

SECONDARY OUTCOMES:
Unilateral isometric adduction strength | Change from baseline isometric adductor strength at 8 weeks
  The player is placed supine and stabilized themselves by holding onto the sides of the examination bed. A belt placed around the pelvis provides further stabilisation. The non-tested leg is placed with knee and hip flexed and the foot flat against the bed. The medial malleolus is in line with the contralateral knee joint line and the toes rest at the end of the bed. The examiner places the HHD 5cm above the medial malleolus and the elbow against the wall for stabilization. Τhe player performs a 5-second MVIC with the instruction to push "as hard as possible". The procedure is repeated two more times with a 30-second rest between each of them and the highest value is recorded.
Delayed onset muscle soreness | Difference in mean muscle soreness at 8 weeks
  Numerical ranking scale from 0 to 10, where 0 is minimum and indicates no muscle soreness, and 10 is maximum and indicates worst imaginable muscle soreness

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Korakakis, PhD, Study Director — Aspetar Orthopaedic & Sports Medicine Hospital
Locations (1):
- Elite football clubs, Athens, Greece

IPD SHARING:
Plan to Share IPD: No